CLINICAL TRIAL: NCT03740633
Title: The Effects of Post-operative Functional Training on the Prevention of Deep Venous Thrombosis in the Patients of Gynecological Malignancies: A Phase 3 Randomized Control Study
Brief Title: Functional Training for the Prevention of Deep Venous Thrombosis
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: Lei Li (Other)
Responsible Party: Sponsor-Investigator, Lei Li, Professor, Peking Union Medical College Hospital
Organization: Peking Union Medical College Hospital (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: GO-FUN
Record Dates: First submitted 2018-11-10; First posted 2018-11-14 (Actual); Last update posted 2018-11-14 (Actual); Status verified 2018-11

CONDITIONS: Ankle Motion; Gynecologic Neoplasm; Deep Venous Thrombosis; Abdominal Breathing
MeSH Terms: conditions — Genital Neoplasms, Female; Venous Thrombosis

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Study group (Experimental): Patients in the study group accept functional training and regular care.
  Interventions: Behavioral: passive ankle pump motions on the day of surgery; Behavioral: active ankle pump motions and abdominal breathing training on the 1-3 day after the surgery; Combination Product: Regular care
- Control group (Active Comparator): Patients in the control group only accept regular care.
  Interventions: Combination Product: Regular care

INTERVENTIONS:
Behavioral: passive ankle pump motions on the day of surgery — Passive ankle pump motions include flexion and extension, circumduction, which will be conducted by caregiver on the day of surgery.
  Arms: Study group
Behavioral: active ankle pump motions and abdominal breathing training on the 1-3 day after the surgery — Active ankle pump motions include flexion and extension, circumduction, which will be conducted by patient on the 1-3 day after the surgery. On the same time, the patient is given abdominal breathing training.
  Arms: Study group
Combination Product: Regular care — Regular post-operative care consists of compression stockings, anticoagulant and instructions of early mobilization

SUMMARY:
This study aims to analyze the post-operative functional training on the prevention of deep venous thrombosis (DVT) in the patients who have accepted major surgeries for the gynecological malignancies. The functional training consists of: (1) active and passive ankle pump motions including flexion and extension, circumduction; (2) abdominal breathing training. The primary end is the incidence of DVT happened 30 days from surgery. The secondary ends include the patients satisfaction about functional training.

ELIGIBILITY:
Inclusion Criteria:

* Having received major surgeries for gynecologic malignancies
* Good performance status
* Aged 18 years or older
* Signed an approved informed consents
* No injuries to the skin, musculoskeletal system
* No venous thromboembolic disease before surgeries

Exclusion Criteria:

* Not meeting all of the inclusion criteria
* Delayed extubation

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 398 (Estimated)
Dates: Start 2018-11-10 (Actual); Primary Completion 2019-11-10 (Estimated); Study Completion 2019-11-10 (Estimated)

PRIMARY OUTCOMES:
deep venous thrombosis | One years
  incidence of deep venous thrombosis

SECONDARY OUTCOMES:
adverse events | One year
  adverse events related to the functional training
patient satisfaction | One year
  patient satisfaction surveyed by customed questionnaire

CONTACTS AND LOCATIONS:
Overall Officials: Lei Li, M.D., Principal Investigator — Peking Union Medical College Hospital
Locations (1):
- Lei Li, Beijing, Beijing Municipality, China